CLINICAL TRIAL: NCT04874597
Title: The Effect of Ocrelizumab on the Peripheral Lymphocyte Immunophenotypes with Suppressive Capacity in Patients with Multiple Sclerosis Previously Treated with Disease Modifying Therapy - a Prospective Exploratory Observational Study
Brief Title: Investigation of the Effect of Ocrelizumab on Peripheral Lymphocyte Immunophenotypes with Suppressive Capacity in MS
Status: Active, not recruiting | Type: Observational
Sponsor: Dr Recai Turkoglu (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr Recai Turkoglu, Principal Investigator, Prof, Haydarpasa Numune Training and Research Hospital
Organization: Haydarpasa Numune Training and Research Hospital (Other)
Other Study IDs: ML42254
Record Dates: First submitted 2021-04-14; First posted 2021-05-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Ocrelizumab; Disease modifying therapy; T cell; B cell
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab treatment will be administered in accordance with the product characteristics approved in Turkey.

SUMMARY:
This is a 24-month, prospective, exploratory, observational study to investigate immune phenotypes in patients with MS following treatment with ocrelizumab.

DETAILED DESCRIPTION:
This is a 24-month, prospective, exploratory, observational study to investigate immune phenotypes in patients with MS following treatment with ocrelizumab. The study will be conducted on Health Sciences University Istanbul Haydarpaşa Numune Training and Research Hospital, Neurology Department.

The decision to treat with ocrelizumab must be made prior to and independently from the proposal to enroll the patient into this study and in line with the Summary of Product Characteristics (SmPC) approved by the Turkish Ministry of Health.

Data will be recorded at screening visit, baseline visit (month 0), second visit on 6th month, third visit on 12th month and last visit (end of the study [EOS]) on 24th month according to local clinic practice. Optional ad hoc visits could be conducted if relapse of MS or infection after vaccination occurs during ocrelizumab treatment.

The duration of the study for each patient will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with a diagnosis of relapsing forms of multiple sclerosis (RMS) or primary progressive multiple sclerosis (PPMS) according to the 2017 revised McDonald criteria.
* Previous MS treatment with at least one of other DMT(*). The patients can be without treatment before switching until the end of wash-out period of previous DMT(s) or until lymphocytes parameter is in normal range.
* Previous treatment change with the reasons inefficacy, safety related issues or lack of compliance.
* Decision to initiate ocrelizumab therapy (in accordance with the product characteristics approved in Turkey) has already been taken for the treatment of MS patient as part of routine clinical practice. The decision to treat with Ocrelizumab must be made prior to and independently from the proposal to enroll the patient into this study.
* Agreed and signed informed consent.

(*) A DMT is defined as any of the following drugs: Teriflunomide, Interferon beta 1a, Interferon beta 1b, Peginterferon beta 1a, Glatiramer acetate, Fingolimod, Daclizumab, Alemtuzumab, Cladribine, Dimethyl fumarate, and Natalizumab.

Exclusion Criteria:

* Previously treated with anti-CD20 therapy (rituximab, atacicept, belimumab or ofatumumab).
* Medical history of a malignancy, active infection (including Hepatitis B virus) or chronic inflammatory disease.
* Medical history or use of any medication other than a DMT as defined above which may affect immunophenotypes of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — MS patients will be stratified for gender to reflect epidemiological incidence of MS subtypes. Gender ratios (Female/Male) for RMS and PPMS are set for 2:1 and 1:1, respectively.
Study Population: A total of 20 MS patients who were previously treated with at least one of other DMT will be recruited. Participants will be recruited by specialized physicians who are experienced in the diagnosis and treatment of MS and ocrelizumab use.
  * Consecutive MS patients with an already planned ocrelizumab therapy will be screened for recruitment in study recruiting clinics. Ocrelizumab treatment will not be initiated to recruit study patients.
  * MS patients will be stratified for gender to reflect epidemiological incidence of MS subtypes. Gender ratios (Female/Male) for RMS and PPMS are set for 2:1 and 1:1, respectively.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in T cell capacity achieved by eliminating B cells as measured by flow cytometry. | From baseline to month 6 and month 12
  Change will be measured in absolute cell numbers and percentages from baseline to Month 6 and to Month 12.
Change from baseline in T cell function achieved by eliminating B cells as measured by flow cytometry. | From baseline to month 6 and month 12
  Change will be measured in absolute cell numbers and percentages from baseline to Month 6 and to Month 12.

SECONDARY OUTCOMES:
Correlation between changes in T and B cell capacity and function during course of ocrelizumab therapy. | Baseline (month 0), month 6 and month 12
Clinical improvement | Baseline (month 0), month 6 and month 12
  Clinical improvement will be confirmed if an increase of less than half a step on the Expanded Disability Status Scale and less than one attack were observed during the first 12 months of ocrelizumab treatment.
Changes in T cells in case of relapse or infection after vaccination during ocrelizumab treatment by flow cytometry. | From baseline (month 0) to month 6 and month 12
Changes in B cells in case of relapse or infection after vaccination during ocrelizumab treatment by flow cytometry. | From baseline (month 0) to month 6 and month 12

OTHER OUTCOMES:
Socio-demographic data | Baseline (month 0)
  Date of birth, sex, country of birth
Previous MS treatment history: DMT agents and other treatments used for MS before ocrelizumab initiation | Screening or baseline (month 0)
  Number (%) patients receiving any DMT agents and other treatments
Previous MS treatment history: dosing, route, and treatment duration | Screening or baseline (month 0)
  Treatment duration: Date of first and last administration for first line DMT agent and other medications used for MS before ocrelizumab initiation
Previous MS treatment history: reasons for discontinuation of each previous MS treatment | Screening or baseline (month 0)
  Reasons for discontinuation includes: inefficacy/high disease activity, relapse, adverse event, lack of compliance or other.
Medical history data | Baseline (month 0)
  Medical history data includes: comorbidities, current and prior treatments for diseases other than MS, hospitalization, surgery, allergies, family history and vaccination history within the last five years.
Vital signs | Baseline (month 0), month 6, month 12 and month 24
  • Heart rate
Vital signs | Baseline (month 0), month 6, month 12 and month 24
  • Blood pressure
Vital signs | Baseline (month 0), month 6, month 12 and month 24
  • Body temperature
Vital signs | Baseline (month 0), month 6, month 12 and month 24
  • Respiratory rate
Physical examination | Baseline (month 0), month 6, month 12 and month 24
  • Height
Physical examination | Baseline (month 0), month 6, month 12 and month 24
  • Weight
Physical examination | Baseline (month 0), month 6, month 12 and month 24
  • Body mass index
Physical examination | Baseline (month 0), month 6, month 12 and month 24
  • Complete neurological and physical examination
Covid-19 assessment | Screening, baseline (month 0), month 6, month 12 and month 24
  Covid-19 polymerase chain reaction (PCR) test result (if available)
Covid-19 assessment | Screening, baseline (month 0), month 6, month 12 and month 24
  Treatment (if available)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Expanded Disability Status Scale (EDSS)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Multiple Sclerosis Functional Composite (MSFC)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Symbol Digit Modalities Test (SDMT)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Nine-Hole Peg Test (9-HPT)
MS Assessment: | Baseline (month 0), month 6, month 12 and month 24
  • Timed 25-foot walk test (25-FWT)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Istanbul Haydarpaşa Numune Training and Research Hospital, Neurology Department, Istanbul, Uskudar, Turkey (Türkiye)